CLINICAL TRIAL: NCT01063608
Title: Study of Immune Responses After Vaccination Against Seasonal Influenza Virus and Against Influenza H1N1-v Pandemic Virus in a Clinical Staff (FLU-HOP)
Brief Title: Study of Immune Responses After Vaccination Against Seasonal Influenza Virus and Against Influenza H1N1-v Pandemic Virus in a Medical Staff.
Acronym: FLU-HOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C09-30; 2009-016267-11 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2010-03

CONDITIONS: Influenza A Virus, H1N1 Subtype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-H1N1v Vaccine (Experimental)
  Interventions: Biological: Anti-H1N1v Vaccine

INTERVENTIONS:
Biological: Anti-H1N1v Vaccine — Inclusion of hospital personnel in the context of the anti-H1N1v prophylaxy plan.

SUMMARY:
This project may help to answer several fundamental questions related to public health regarding vaccination against influenza viruses and regarding the influenza A(H1N1)v pandemy:

What is the immunologic efficacy in terms of antibodies response of the vaccination against the seasonal (2009-2010) influenza virus and against the A(H1N1)v virus in the clinical staff?

Moreover, it may help to answer questions related to the use of a vaccine against influenza virus variants emerging in the French population:

1. Before the vaccination:

   * What is the status of the residual anti-H1N1 seasonal viruses immunity and of the anti-A(H1N1)v immunity in the population stratified by age and taking into account the multiplicity of the prior seasonal vaccinations?
   * What is the level of the cellular and humoral cross-reactivity between the different H1N1 strains?
2. After the vaccination:

   * What is the intensity of the anti-vaccine immune response as a function of the age of the population ad of the prior seasonal vaccinations?
   * What is the level of the cellular and humoral cross-reactivity after vaccination as a function of the age of the population and of the multiplicity of the prior seasonal vaccinations?

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age superior or equal to 20 years
* Women with childbearing potential using contraception

Exclusion Criteria:

* Documented immune depression
* Current immunosuppressive therapy
* Pregnancy (documented by a positive pregnancy test)
* Breast feeding women
* Documented allergy or hypersensitivity to vaccines
* Documented acute or chronic inflammatory disease
* Concomitant participation to another clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the intensity of the humoral and cellular immune responses of the anti-A(H1N1)v vaccine in a medical care population as a function of the age and of the prior seasonal anti-influenza vaccinations. | 5 months

SECONDARY OUTCOMES:
Investigate the quality of the humoral and cellular immune responses induced by the seasonal anti-influenza vaccine as a function of the age and of the prior seasonal vaccinations. | 5 months
Determine the cross-reactivity of the humoral and cellular immune responses as a function of the age and of the prior seasonal vaccinations | 5 months
Assess the tolerance to the seasonal and pandemic vaccines | 5 months
Assess the occurence of flu episodes and their severity during the 2009-2010 season as a function of the age of the population. Then, the correlation between the flu episodes and and the immunologic results is to be evaluated. | 5 months
Evaluate the perception of the anti-influenza vaccination in a medical care population in the current H1N1v pandemy context. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Jaureguiberry, MD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière; Behazine Combadiere, PhD, Study Director — INSERM U945
Locations (2):
- France (2):
  - Hopital Pitie Salpetriere, Paris, Île-de-France Region
  - Centre d'Investigations Cliniques (CIC), Hopital Cochin, Paris, Île-de-France Region

REFERENCES:
- [Background] Bonduelle O, Yahia N, Siberil S, Benhabiles N, Carrat F, Krivine A, Rozenberg F, Dimitrov J, Kaveri SV, Curjol A, Tindel M, Louet M, Desert F, Launay O, Loulergue P, Badre G, Katlama C, Bricaire F, Samri A, Rousset D, van der Werf S, Jaureguiberry S, Combadiere B. Longitudinal and integrative biomodeling of effector and memory immune compartments after inactivated influenza vaccination. J Immunol. 2013 Jul 15;191(2):623-31. doi: 10.4049/jimmunol.1203483. Epub 2013 Jun 17. PMID 23776176
- See also: Publication report Results — https://journals.aai.org/jimmunol/article/191/2/623/83692/Longitudinal-and-Integrative-Biomodeling-of